CLINICAL TRIAL: NCT05036408
Title: Cancer Pain Rehabilitation Program in Cancer Survivorship Feasibility Study
Brief Title: Cancer Pain Rehabilitation Program to Reduce Pain Related Distress, and Reliance of Pain Medication Through Multimodal Nonpharmacological Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19530; NCI-2021-02052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19530 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-07-01; First posted 2021-09-05 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Occupational Therapy; Exercise; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (cancer pain rehabilitation program) (Experimental): Patients participate in the cancer pain rehabilitation program for 6 weeks, including educational sessions over 2 hours once weekly, group psychological interventions, group physical therapy, and 1:1 physical and occupational therapy treatment per the patient's treatment plan. Patients may also undergo osteopathic manual treatments per physical and occupational therapy assessments.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Educational Intervention; Procedure: Manipulative and Body-Based Intervention Procedure; Behavioral: Occupational Therapy; Other: Physical Activity; Procedure: Physical Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Participate in group psychological intervention
Other: Educational Intervention — Attend educational session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Procedure: Manipulative and Body-Based Intervention Procedure — Undergo osteopathic manual treatments
  Other Names: Manipulative and Body-Based Intervention; Manipulative and Body-Based Methods; Manipulative and Body-Based Systems
Behavioral: Occupational Therapy — Participate in occupational therapy
  Other Names: OT
Other: Physical Activity — Participate in physical activity
Procedure: Physical Therapy — Participate in physical therapy
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect of an interdisciplinary program with strong patient involvement on managing long-term chronic pain for cancer survivors. The purpose of this study is to determine whether enrolling patients into an interdisciplinary program can improve mobility with physical and occupational therapy and participation in online group psychotherapy that teaches coping skills to enhance quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To test the feasibility of an interdisciplinary functional restoration program in cancer survivors with chronic pain and restoring physical function.

EXPLORATORY OBJECTIVE:

I. To explore the preliminary effect of functional restoration program (FRP) in restoring physical function and reducing pain which ultimately decreases opioid consumption.

OUTLINE:

Patients participate in the cancer pain rehabilitation program for 6 weeks, including educational sessions over 2 hours once weekly, group psychological interventions, group physical therapy, and 1:1 physical and occupational therapy treatment per the patient's treatment plan. Patients may also undergo osteopathic manual treatments per physical and occupational therapy assessments.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted in those with history of cancer in remission or with stable disease living with chronic pain greater than 6 months in duration
* Cancer survivors or stable indolent cancer patients ages 18 or older living with chronic pain
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients are required to have access to a computer with a camera and a reliable internet connection. The education lectures and psychotherapy group components of the program are facilitated via online Health Insurance Portability and Accountability Act (HIPPA) compliant platform
* Eligible participants will be able to read and write and speak English and be motivated and able to commit to attending six consecutive weekly group and individual sessions

Exclusion Criteria:

* Patients who are less than the age of 18 or have active problems with addiction will be excluded:

  * Those identified with illicit substance abuse or addiction will be referred to an addiction specialist or medication assisted treatment program through our resource coordinator
  * "Active substance abuse" exclusion was defined using the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) Criteria which is the gold standard for diagnosing substance use disorders is a cluster of cognitive, behavioral and physiological symptoms indicated that the individual continues using the substance despite significant substance related problems
  * The substances that were considered are listed below:

    * Alcohol
    * Cannabis
    * Hallucinogens
    * Inhalants
    * Opioids
    * Sedatives (hypnotics or anxiolytics)
    * Stimulants
  * Overall, the diagnosis was based on pathological patterns of behaviors related to the use of the substance. Criteria that fit with overall groupings include impaired control, social impairment, risky use, and pharmacological criteria
* Impaired control

  * The individual may express overall desire to cut down or regulate substance use and may report multiple unsuccessful efforts to decrease or discontinue use
  * The individual may spend a great deal of time obtaining the substance, using the substance, or recovering from its affects
  * The individual's daily activities revolve around the substance in some instances of more severe substance use disorder
  * Craving is manifested by intense desire or urge for the drug that may occur at any time
* Social impairment

  * Recurrent substance use may result in failure to fulfill major role obligations at work, school, or home
  * The individual may continue substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance
  * Important social, occupational, or recreational activities may be given up or reduced because of substance use
  * The individual may withdraw from family activities and hobbies in order to use the substance
* Risky use

  * Recurrent use in situations in which it is physically hazardous
  * The individual may continue substance use despite knowledge of having persistent or recurrent physical or psychological problem that is likely to have been caused or exacerbated by the substance
* Pharmacologic criteria

  * Tolerance is signaled by requiring a markedly increased dose of substance to achieve the desired effect or markedly reduced effect when the usual dose is consumed
  * Withdrawal is a syndrome that occurs when blood or tissue concentrations of a substance decline in an individual who had maintained a prolonged heavy use of the substance
  * After developing withdrawal symptoms, the individual is likely to consume the substance to relieve the symptoms

    * Symptoms of tolerance or withdrawal occurring during appropriate medication treatment with prescribed medications are specifically not counted. However, prescription medications can be used inappropriately based on criteria above and substance use disorder can be correctly diagnosed when there are other symptoms of compulsive and drug seeking behavior
* Substance use disorders occur in a broad range of severity from mild to severe with severity based on number of symptom criteria endorsed.

  * Mild

    * Presence of 2-3 symptoms
  * Moderate

    * Presence of 4-5 symptoms
  * Severe

    * Presence of 6-7 symptoms
* For our research purposes, our exclusion criteria included any individual who met criteria for mild, moderate, and severe substance use disorder
* Those with severe cognitive or psychiatric impairments that preclude participation in group sessions will be excluded
* Patients should not have any uncontrolled illness of any kind including ongoing or active infection
* Subjects, who are not be able to comply with the safety monitoring requirements of the study. Those who miss more than half the sessions will be considered to not have completed the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of Functional Restoration Program | 24 months from the intervention date
  Feasibility of the program will be determined by the proportion of referred eligible cancer survivors enrolled into the program (at least 50% who are eligible enroll) and the proportion of enrolled patients completed at least half of the intervention.

OTHER OUTCOMES:
Preliminary effect of the Functional Restoration Program in reducing pain (NSR) | Pre-intervention , End of intervention (6 weeks), 3 months post-intervention
  Pain Numerical Rating Scale (NSR) score: patients are asked to circle the number between 0 and 10, zero usually represents 'no pain at all' whereas the upper limit 10 represents 'the worst pain ever possible'.
Preliminary effect of the Functional Restoration Program in reducing pain (PSEQ) | Pre-intervention, End of intervention (6 weeks), 3 months post-intervention
  The Pain Self-Efficacy Questionnaire (PSEQ) score: the PSEQ is a 10-item questionnaire, developed to assess the confidence people with ongoing pain have in performing activities while in pain. Scores can range from 0 - 60 and is done by simple addition. High PSEQ scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients. Higher scores (and a higher percentile) represent lower confidence to function with pain.
Preliminary effect of the Functional Restoration Program to restore physical function (ADL) | Pre-intervention, End of intervention (6 weeks), 3 months post-intervention
  Activities of Daily Living (ADL): Medical Outcomes Study [MOS] subscale, Measures limitations in physical function activities, ranging from bathing and dressing to running.
Preliminary effect of the Functional Restoration Program to restore physical function (OARS) | Pre-intervention, End of intervention (6weeks), 3 months post-intervention
  Instrumental Activities of Daily Living (iADL): Older American Resources and Services [OARS] subscale, Measures ability to complete activities required to maintain independence, ranging from making telephone calls to money management.
Preliminary effect of the Functional Restoration Program to restore physical function (6MWT) | Pre-intervention, End of intervention (6 weeks), 3 months post-intervention
  Six minutes walk test (6MWT): The 6-min walk test is a submaximal exercise test that entails the measurement of distance (meter) walked over a span of 6 minutes.
Preliminary effect of the Functional Restoration Program to restore physical function (10mWT) | Pre-intervention, End of intervention (6 weeks), 3 months post-intervention
  Ten meter walking test (10mWT): The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.

CONTACTS AND LOCATIONS:
Overall Officials: Heather N Bitar, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States